CLINICAL TRIAL: NCT01965288
Title: A Single-Center Study Comparing the Clinical Performance of Biofinity Toric Versus Air Optix for Astigmatism Over 1 Month of Daily Wear.
Brief Title: Clinical Performance of Biofinity Toric Versus Air Optix for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-42
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A (Experimental): Each subject randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating the schedule for the second pair without a washout period.
  Interventions: Device: comfilcon A; Device: lotrafilcon B
- lotrafilcon B (Active Comparator): Each subject randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating the schedule for the second pair without a washout period.
  Interventions: Device: comfilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: comfilcon A — test lens Pair(comfilcon A) or the control lens Pair(lotrafilcon B)
  Other Names: Biofinity Toric
Device: lotrafilcon B — test lens Pair(comfilcon A) or the control lens Pair(lotrafilcon B)
  Other Names: Air Optix

SUMMARY:
The aim of this study is to compare the clinical performance of the Biofinity Toric (comfilcon A) contact lens, versus Air Optix for Astigmatism (lotrafilcon B) over 1 month of daily wear.

DETAILED DESCRIPTION:
Single masked, open label, randomized, bilateral, crossover study design comparing comfilcon A against lotrafilcon B lenses over 1 month of daily wear for each study lens. Each subject will be randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating the schedule for the second pair without a washout period.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft toric contact lens wearer
* Has a contact lens spherical prescription between +6.00 to - 10.00 (inclusive)
* Have no less than 0.75diopter (D) of astigmatism and no more than 2.25D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a contact lens prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.25 D of cylinder in either eye.
* Has a history of not achieving comfortable contact lens wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, OD MPhil PhD, Principal Investigator — Optometry Research Group (GIO) - Optics Department, University of Valencia
Locations (1):
- Optometry Research Group (GIO) - Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 60 subjects enrolled, 60 were fitted with the study lenses and completed the trial (i.e.
  no discontinuations).This study design considered a single-center, (Optometry Research Group), located at the University of Valencia Spain (target 60 subjects).
Pre-assignment Details: All subjects were habitual lens wearers.
Groups:
- Comfilcon A Then Lotrafilcon B; Lotrafilcon B Then Comfilcon A: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
Period: Overall Study
Arm/Group | Comfilcon A Then Lotrafilcon B | Lotrafilcon B Then Comfilcon A
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The subject sample consisted of sixty (60) habitual toric contact lens wearers.
Groups:
- Comfilcon A Then Lotrafilcon B; Lotrafilcon B Then Comfilcon A: All subjects attended first visit with habitual lenses and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
- Total: Total of all reporting groups
Arm/Group | Comfilcon A Then Lotrafilcon B | Lotrafilcon B Then Comfilcon A | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 14 | 9 | 23
Region of Enrollment [Number; unit: participants]
  Spain | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Daily and Comfortable Wearing Time
Description: Participant rating of lens Daily and Comfortable Wearing Time. Collected at baseline for all habitual lenses. (The hours of average comfortable wearing time and average daily wearing time.)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Overall Study Group: All 60 subjects wearing habitual lens prior to dispense of study lens.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
hours
  Average comfortable wearing time | 8.8 (2.5)
  Average daily wearing time | 9.2 (2.6)

2. Secondary Outcome: Limbal Hyperaemia
Description: Assessment of ocular health. Collected at baseline after removal of habitual lenses. Proportion of eyes with grades 0-1 (No eyes graded >1) (Biomicroscopy, 0-4, ½ grades; 0=none: no injection present, 4=severe)
Time Frame: Baseline
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Overall Study Group: All 60 subjects after removal of habitual lens and prior to dispense of study lens.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 97.5
  Grade 1/2 | 2.5
  Grade 1 | 0.0

3. Primary Outcome: Comfort, Dryness, Handling, Lens Fit Stability, Vision Satisfaction
Description: Participant rating of lens Comfort, Dryness, Handling, Lens Fit Stability and Vision Satisfaction. Collected at baseline for all habitual lenses. (0-10; Comfort, Lens Fit and Satisfaction / 0=very poor,10=excellent; Dryness / 0=very dry, 10=no dryness; Handling / 0=very difficult, 10=very easy for handling)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
units on a scale
  Comfort on Insertion | 8.0 (1.3)
  Comfort prior to Removal | 7.7 (1.6)
  Comfort Overall | 8.0 (1.6)
  Dryness during the Day | 8.0 (1.6)
  Dryness prior to Removal | 7.9 (1.6)
  Dryness Overall | 7.9 (1.6)
  Handling | 8.4 (1.1)
  Overall Lens Fit | 8.2 (1.1)
  Overall Vision Satisfaction | 8.1 (1.2)

4. Primary Outcome: Vision Quality Insertion, During Day, End Day
Description: Participant rating of vision quality on insertion, during the day, end of day. Collected at baseline for all habitual lenses. (0-100; 0=extremely poor vision totally blurred, 100=excellent vision totally sharp)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
units on a scale
  On Insertion | 78.5 (12.4)
  During the Day | 82.7 (13.2)
  End of Day | 80.2 (14.3)

5. Primary Outcome: Vision Stability Insertion, During Day, End Day
Description: Participant rating of vision stability on insertion, during the day, end of day. Collected at baseline for all habitual lenses. (0-100; 0=totally unstable fluctuating/changing, 100=perfectly stable not fluctuating/changing)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
units on a scale
  On Insertion | 78.5 (12.0)
  During the Day | 83.8 (13.4)
  End of Day | 82.9 (13.3)

6. Primary Outcome: Overall Sensation of Moistness
Description: Participant rating for overall sensation of moistness. Collected at baseline for all habitual lenses. (5-point Likert Scale; Excellent, Good, Average, Below Average)
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of subjects
  Excellent | 23
  Good | 25
  Average | 50
  Below Average | 0
  Poor | 2

7. Primary Outcome: Overall Sensation of Smoothness
Description: Participant rating for overall sensation of smoothness. Collected at baseline for all habitual lenses. (5-point Likert Scale; Excellent, Good, Average, Below Average)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Excellent | 27
  Good | 33
  Average | 40
  Below Average | 0
  Poor | 0

8. Primary Outcome: Comfort Satisfaction
Description: Participant rating for comfort satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 37
  Somewhat Satisfied | 55
  Somewhat Dissatisfied | 7
  Completely Dissatisfied | 2

9. Primary Outcome: Dryness Satisfaction
Description: Participant rating for dryness satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 33
  Somewhat Satisfied | 53
  Somewhat Dissatisfied | 12
  Completely Dissatisfied | 2

10. Primary Outcome: Handling Satisfaction
Description: Participant rating for handling satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 57
  Somewhat Satisfied | 37
  Somewhat Dissatisfied | 5
  Completely Dissatisfied | 2

11. Primary Outcome: Lens Fit Satisfaction
Description: Participant rating for lens fit satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 42
  Somewhat Satisfied | 50
  Somewhat Dissatisfied | 8
  Completely Dissatisfied | 0

12. Primary Outcome: Vision Satisfaction
Description: Participant rating for vision satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 48
  Somewhat Satisfied | 45
  Somewhat Dissatisfied | 7
  Completely Dissatisfied | 0

13. Primary Outcome: Overall Satisfaction
Description: Participant rating for overall satisfaction. Collected at baseline for all habitual lenses. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
percentage of participants
  Completely Satisfied | 40
  Somewhat Satisfied | 53
  Somewhat Dissatisfied | 7
  Completely Dissatisfied | 0

14. Primary Outcome: Comfort Upon Contact Lens Insertion
Description: Participant rating of comfort upon insertion. Collected at dispense for each lens. (0-10; 10=Can't Feel)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A; Lotrafilcon B: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale | 9.0 (0.8) | 7.8 (1.2)

15. Primary Outcome: Vision Satisfaction Upon Contact Lens Insertion
Description: Participant rating of vision satisfaction upon insertion. Collected at dispense for each lens. (0-10; 10= Very Satisfied)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale | 8.8 (1.1) | 8.2 (1.3)

16. Primary Outcome: Vision Quality With Contact Lens Prescription
Description: Participant rating of Vision Quality with contact lens prescription. Collected at dispense for each lens. (0-100; 0=extremely poor vision totally blurred, 100=excellent vision totally sharp)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale | 88 (9.3) | 82 (11.9)

17. Primary Outcome: Vision Stability Upon Contact Lens Insertion
Description: Participant rating of vision stability on insertion. Collected at dispense for each lens. (0-100; 0=extremely poor vision totally blurred, 100=excellent vision totally sharp)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale | 87 (11.9) | 82 (11.7)

18. Primary Outcome: Visual Acuity logMAR
Description: Assessment of monocular and binocular high and low contrast visual acuity (VA). Collected at dispense for each lens. logMAR (VA).
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Log Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
logMAR
  MHCVA (OU Average) | -0.02 (0.05) | -0.01 (0.06)
  MLCVA (OU Average) | 0.18 (0.05) | 0.19 (0.07)
  BHCVA | -0.04 (0.06) | -0.02 (0.05)
  BLCVA | 0.17 (0.07) | 0.18 (0.05)

19. Primary Outcome: Centration
Description: Assessment of Lens Fit Performance for centration. Collected at dispense for each lens. (Biomicroscopy; centered or slightly decentered)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  centered | 94 | 79
  slightly decentered | 6 | 21

20. Primary Outcome: Corneal Coverage
Description: Assessment of Lens Fit Performance for corneal coverage. Collected at dispense for each lens. Corneal coverage assessed in primary gaze: (yes=full corneal coverage at all times, no=incomplete corneal coverage)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses | 100 | 100

21. Primary Outcome: Post Blink Movement
Description: Assessment of Lens Fit Performance for post blink movement. Collected at dispense for each lens. (0-4, 0.5 increments; 0=Insufficient, unacceptable movement, 4= Excessive, unacceptable movement)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
units on a scale | 0.09 (0.30) | 0.19 (0.42)

22. Primary Outcome: Lens Orientation Primary Gaze
Description: Assessment of Lens Fit Performance for lens orientation in primary position of gaze. Collected at dispense for each lens. (Degree of mislocation relative to lens axis mark.)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
degrees | 0.71 (1.75) | 1.06 (1.90)

23. Primary Outcome: Lens Marking Visibility
Description: Assessment of Lens Fit Performance for lens marking visibility. Collected at dispense for each lens. (1-3, 1=excellent, 2=average, 3=poor)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Excellent | 89 | 42
  Average | 11 | 42
  Poor | 0 | 16

24. Primary Outcome: Lens Stability on Blink
Description: Assessment of Lens Fit Performance for lens rotational stability on blink. Collected at dispense for each lens. (No rotation and 5-10 degrees rotation from axis location mark)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  No rotation | 100 | 98
  5-10 degrees | 0 | 2

25. Primary Outcome: Lens Stability 5-10 Min
Description: Assessment of Lens Fit Performance for lens to stabilize in 5-10 min. Collected at dispense for each lens. (Varied less than 5 degrees from lens marking location between 5-10 min)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses | 100 | 100

26. Primary Outcome: Lens Overall Stability
Description: Assessment of Lens Fit Performance for overall lens stability. Collected at dispense for each lens. (Excellent or Good)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Excellent | 80 | 50
  Good | 20 | 50

27. Primary Outcome: Rotational Recovery 30/45 Deg
Description: Assessment of Lens Fit Performance for lens rotational recovery to original position. Collected at dispense for each lens. Assessed in degree of mislocation relative to original position after manual temporal rotation. (30 deg/10 blinks, 45 deg/60 sec)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
degrees
  30 deg/ 10 blinks | 0.542 (1.56) | 0.833 (1.98)
  45 deg/ 60 sec | 0.625 (1.66) | 0.875 (2.01)

28. Primary Outcome: Overall Fit Acceptance
Description: Assessment of Lens Fit Performance for overall lens fit acceptance. Collected at dispense for each lens. Rated perfect or not perfect based on lens fit alone. (0-4; 0=should not be worn, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: Dispense
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses fitted
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses fitted
  Perfect | 82 | 57
  Not Perfect | 18 | 43

29. Primary Outcome: Daily and Comfortable Wearing Time
Description: Participant rating of lens Daily and Comfortable Wearing Time. Collected at 2 weeks wear for each lens. (The hours of average comfortable wearing time and average daily wearing time.)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
hours
  average comfortable wearing time | 9.8 (2.3) | 8.3 (3.0)
  average daily wearing time | 10.1 (2.0) | 10.1 (1.8)

30. Primary Outcome: Daily and Comfortable Wearing Time
Description: Participant rating of lens Daily and Comfortable Wearing Time. Collected at 4 weeks wear for each lens. (The hours of average comfortable wearing time and average daily wearing time.)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
hours
  average comfortable wearing time | 9.5 (2.1) | 7.8 (2.8)
  average daily wearing time | 9.9 (1.7) | 9.8 (1.7)

31. Primary Outcome: Participants Use of Rewetting Drops
Description: Proportion of subjects using rewetting drops. Collected at 2 weeks for each lens. (Yes, No)
Time Frame: 2 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants | 7 | 50

32. Primary Outcome: Participants Use of Rewetting Drops
Description: Proportion of subjects using rewetting drops. Collected at 4 weeks for each lens. (Yes, No)
Time Frame: 4 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants | 15 | 58

33. Primary Outcome: Comfort, Dryness, Handling, Lens Fit Stability, Vision Satisfaction
Description: Participant rating of lens Comfort, Dryness, Handling, Lens Fit Stability and Vision Satisfaction. Collected at 2 weeks wear for each lens. (0-10; Comfort, Lens Fit and Satisfaction / 0=very poor,10=excellent; Dryness / 0=very dry, 10=no dryness; Handling / 0=very difficult, 10=very easy for handling)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  Comfort on Insertion | 8.7 (1.1) | 7.7 (1.3)
  Comfort prior to Removal | 8.7 (1.1) | 7.4 (1.4)
  Comfort Overall | 8.8 (1.1) | 7.6 (1.3)
  Dryness during the Day | 8.7 (1.3) | 7.6 (1.4)
  Dryness prior to Removal | 8.6 (1.5) | 7.5 (1.5)
  Dryness Overall | 8.7 (1.3) | 7.5 (1.5)
  Handling | 8.3 (1.1) | 8.0 (1.6)
  Lens Fit Stability | 8.8 (1.2) | 8.0 (1.5)
  Vision Satisfaction | 8.7 (1.1) | 8.0 (1.5)

34. Primary Outcome: Comfort, Dryness, Handling, Lens Fit Stability, Vision Satisfaction
Description: Participant rating of lens Comfort, Dryness, Handling, Lens Fit Stability and Vision Satisfaction. Collected at 4 weeks wear for each lens. (0-10; Comfort, Lens Fit and Satisfaction / 0=very poor,10=excellent; Dryness / 0=very dry, 10=no dryness; Handling / 0=very difficult, 10=very easy for handling)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  Comfort on Insertion | 8.6 (1.0) | 7.1 (1.5)
  Comfort prior to Removal | 8.5 (1.1) | 6.7 (1.6)
  Comfort Overall | 8.6 (1.1) | 6.9 (1.6)
  Dryness during the Day | 8.5 (1.1) | 7.0 (1.6)
  Dryness prior to Removal | 8.5 (1.1) | 7.0 (1.5)
  Dryness Overall | 8.6 (1.1) | 7.0 (1.6)
  Handling | 8.2 (1.1) | 7.8 (1.7)
  Lens Fit Stability | 8.6 (1.1) | 7.6 (1.6)
  Vision Satisfaction | 8.5 (1.0) | 7.6 (1.6)

35. Primary Outcome: Vision Quality Insertion, During Day, End Day, Night
Description: Participant rating of vision quality on insertion, during the day, end of day and night. Collected at 2 weeks wear for each lens. (0-100; 0=extremely poor vision totally blurred, 100=excellent vision totally sharp)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lotrafilcon B: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.)
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  On Insertion | 88 (8) | 84 (9)
  During the Day | 89 (9) | 85 (10)
  End of Day | 87 (9) | 83 (11)
  Night | 84 (9) | 80 (12)

36. Primary Outcome: Vision Quality Insertion, During Day, End Day, Night
Description: Participant rating of vision quality on insertion, during the day, end of day and night. Collected at 4 weeks wear for each lens. (0-100; 0=extremely poor vision totally blurred, 100=excellent vision totally sharp)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  On Insertion | 85 (10) | 79 (11)
  During the Day | 88 (10) | 82 (13)
  End of Day | 86 (11) | 80 (13)
  Night | 83 (10) | 76 (12)

37. Primary Outcome: Vision Stability on Insertion, During Day, End Day
Description: Participant rating of vision stability on insertion, during the day, end of day. Collected at 2 weeks wear for each lens. (0-100; 0=totally unstable fluctuating/changing, 100=perfectly stable not fluctuating/changing)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.A)
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  On Insertion | 87 (9) | 83 (11)
  During the Day | 91 (9) | 85 (13)
  End of Day | 89 (10) | 84 (12)

38. Primary Outcome: Vision Stability on Insertion, During Day, End Day
Description: Participant rating of vision stability on insertion, during the day, end of day. Collected at 4 weeks wear for each lens. (0-100; 0=totally unstable fluctuating/changing, 100=perfectly stable not fluctuating/changing)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
units on a scale
  On Insertion | 85 (10) | 80 (13)
  During the Day | 87 (11) | 82 (14)
  End of Day | 86 (9) | 80 (13)

39. Primary Outcome: Overall Sensation of Moistness
Description: Participant rating for overall sensation of moistness. Collected at 2 weeks wear for each lens. (5-point Likert Scale; Excellent, Good, Average, Below Average, Poor)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Excellent | 57 | 20
  Good | 30 | 30
  Average | 13 | 33
  Below Average | 0 | 12
  Poor | 0 | 5

40. Primary Outcome: Overall Sensation of Moistness
Description: Participant rating for overall sensation of moistness. Collected at 4 weeks wear for each lens. (5-point Likert Scale; Excellent, Good, Average, Below Average, Poor)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Excellent | 60 | 18
  Good | 27 | 23
  Average | 12 | 30
  Below Average | 2 | 25
  Poor | 0 | 3

41. Primary Outcome: Overall Sensation of Smoothness
Description: Participant rating for overall sensation of smoothness. Collected at 2 weeks wear for each lens. (5-point Likert Scale; Excellent, Good, Average, Below Average, Poor)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Excellent | 48 | 27
  Good | 38 | 30
  Average | 13 | 30
  Below Average | 0 | 12
  Poor | 0 | 2

42. Primary Outcome: Overall Sensation of Smoothness
Description: Participant rating for overall sensation of smoothness. Collected at 4 weeks wear for each lens. (5-point Likert Scale; Excellent, Good, Average, Below Average, Poor)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Excellent | 47 | 13
  Good | 42 | 38
  Average | 10 | 28
  Below Average | 2 | 17
  Poor | 0 | 3

43. Primary Outcome: Comfort Satisfaction
Description: Participant rating for comfort satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 72 | 25
  Somewhat Satisfied | 23 | 45
  Somewhat Dissatisfied | 5 | 28
  Completely Dissatisfied | 0 | 2

44. Primary Outcome: Comfort Satisfaction
Description: Participant rating for comfort satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 72 | 27
  Somewhat Satisfied | 23 | 37
  Somewhat Dissatisfied | 5 | 27
  Completely Dissatisfied | 0 | 10

45. Primary Outcome: Dryness Satisfaction
Description: Participant rating for dryness satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 73 | 32
  Somewhat Satisfied | 27 | 42
  Somewhat Dissatisfied | 0 | 25
  Completely Dissatisfied | 0 | 1.7

46. Primary Outcome: Dryness Satisfaction
Description: Participant rating for dryness satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 77 | 23
  Somewhat Satisfied | 13 | 35
  Somewhat Dissatisfied | 10 | 32
  Completely Dissatisfied | 0 | 10

47. Primary Outcome: Handling Satisfaction
Description: Participant rating for handling satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 47 | 45
  Somewhat Satisfied | 42 | 43
  Somewhat Dissatisfied | 12 | 10
  Completely Dissatisfied | 0 | 1.7

48. Primary Outcome: Handling Satisfaction
Description: Participant rating for handling satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 42 | 40
  Somewhat Satisfied | 48 | 48
  Somewhat Dissatisfied | 10 | 12
  Completely Dissatisfied | 0 | 0

49. Primary Outcome: Vision Satisfaction
Description: Participant rating for vision satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 70 | 43
  Somewhat Satisfied | 30 | 48
  Somewhat Dissatisfied | 0 | 7
  Completely Dissatisfied | 0 | 2

50. Primary Outcome: Vision Satisfaction
Description: Participant rating for vision satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 63 | 35
  Somewhat Satisfied | 32 | 53
  Somewhat Dissatisfied | 5 | 12
  Completely Dissatisfied | 0 | 0

51. Primary Outcome: Lens Fit Satisfaction
Description: Participant rating for lens fit satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 70 | 45
  Somewhat Satisfied | 27 | 47
  Somewhat Dissatisfied | 3 | 7
  Completely Dissatisfied | 0 | 2

52. Primary Outcome: Lens Fit Satisfaction
Description: Participant rating for lens fit satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 70 | 35
  Somewhat Satisfied | 25 | 55
  Somewhat Dissatisfied | 5 | 10
  Completely Dissatisfied | 0 | 0

53. Primary Outcome: Overall Satisfaction
Description: Participant rating for overall satisfaction. Collected at 2 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 68 | 30
  Somewhat Satisfied | 30 | 45
  Somewhat Dissatisfied | 2 | 23
  Completely Dissatisfied | 0 | 2

54. Primary Outcome: Overall Satisfaction
Description: Participant rating for overall satisfaction. Collected at 4 weeks wear for each lens. (4-point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Groups:
- Comfilcon A: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.)
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Completely Satisfied | 65 | 22
  Somewhat Satisfied | 28 | 45
  Somewhat Dissatisfied | 7 | 27
  Completely Dissatisfied | 0 | 7

55. Primary Outcome: Wavefront Aberrations Root Mean Square (RMS) (3mm)
Description: Assessment of wavefront aberrations. Collected at 2 weeks for each lens. Wavefront measurement (3mm), Scale in microns (µm).
Time Frame: 2 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
microns
  HOA | 0.065 (0.061) | 0.07 (0.066)
  Third Order | 0.043 (0.054) | 0.046 (0.041)
  Fourth Order | 0.034 (0.049) | 0.029 (0.051)

56. Primary Outcome: Wavefront Aberrations RMS (3mm)
Description: Assessment of wavefront aberrations. Collected at 4 weeks for each lens. Wavefront measurement (3mm), Scale in microns (µm).
Time Frame: 4 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
microns
  HOA | 0.071 (0.052) | 0.075 (0.063)
  Third Order | 0.047 (0.051) | 0.05 (0.048)
  Fourth Order | 0.033 (0.061) | 0.03 (0.059)

57. Primary Outcome: Wavefront Aberrations RMS (5mm)
Description: Assessment of wavefront aberrations. Collected at 2 weeks for each lens. Wavefront measurement (5 mm), Scale in microns (µm).
Time Frame: 2 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
microns
  HOA | 0.214 (0.052) | 0.223 (0.063)
  Third Order | 0.156 (0.041) | 0.161 (0.052)
  Fourth Order | 0.071 (0.031) | 0.075 (0.032)

58. Primary Outcome: Wavefront Aberrations RMS (5mm)
Description: Assessment of wavefront aberrations. Collected at 4 weeks for each lens. Wavefront measurement (5 mm), Scale in microns (µm).
Time Frame: 4 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
microns
  HOA | 0.261 (0.065) | 0.287 (0.075)
  Third Order | 0.161 (0.042) | 0.167 (0.055)
  Fourth Order | 0.075 (0.0291) | 0.081 (0.034)

59. Primary Outcome: Visual Acuity logMAR
Description: Assessment of monocular and binocular high and low contrast visual acuity (VA). Collected at 2 weeks for each lens. logMAR (VA).
  Monocular High Contrast Visual Acuity (MHCVA), Monocular Low Contrast Visual Acuity (MLCVA), Binocular High Contrast Visual Acuity (BHCVA), Binocular Low Contrast Visual Acuity (BLCVA)
Time Frame: 2 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Log Mean (Standard Deviation); unit: logMAR
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
logMAR
  MHCVA (both eyes Average) | -0.01 (0.05) | -0.01 (0.05)
  MLCVA (both eyes Average) | 0.19 (0.05) | 0.19 (0.05)
  BHCVA | -0.04 (0.05) | -0.03 (0.05)
  BLCVA | 0.17 (0.05) | 0.18 (0.05)

60. Primary Outcome: Visual Acuity logMAR
Description: Assessment of monocular and binocular high and low contrast visual acuity (VA). Collected at 4 weeks for each lens. logMAR (VA).
  Monocular High Contrast Visual Acuity (MHCVA), Monocular Low Contrast Visual Acuity (MLCVA), Binocular High Contrast Visual Acuity (BHCVA), Binocular Low Contrast Visual Acuity (BLCVA)
Time Frame: 4 Weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Log Mean (Standard Deviation); unit: logMAR
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
logMAR
  MHCVA (both eyes Average) | -0.01 (0.05) | -0.01 (0.05)
  MLCVA (both eyes Average) | 0.19 (0.05) | 0.19 (0.05)
  BHCVA | -0.03 (0.05) | -0.03 (0.05)
  BLCVA | 0.18 (0.05) | 0.18 (0.05)

61. Primary Outcome: Lens Orientation Primary Gaze
Description: Assessment of Lens Fit Performance for lens orientation in primary position of gaze. Assessed at 2 weeks wear for each lens. (Degree of mislocation relative to lens axis mark.)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
degrees | 0.67 (1.71) | 1.17 (2.22)

62. Primary Outcome: Lens Orientation Primary Gaze
Description: Assessment of Lens Fit Performance for lens orientation in primary position of gaze. Assessed at 4 weeks wear for each lens. (Degree of mislocation relative to lens axis mark.)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
degrees | 0.87 (2.01) | 1.08 (2.17)

63. Primary Outcome: Rotational Recovery 30/45 Deg
Description: Assessment of Lens Fit Performance for lens rotational recovery to original position. Collected at 2 weeks wear for each lens. Assessed in degree of mislocation relative to original position after manual temporal rotation. (30 deg/10 blinks, 45 deg/60 sec)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
degrees
  30 deg/ 10 blinks | 0.25 (1.09) | 0.83 (1.98)
  45 deg/ 60 sec | 0.58 (1.61) | 0.96 (2.08)

64. Primary Outcome: Rotational Recovery 30/45 Deg
Description: as for outcome 63
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
degrees
  30 deg/ 10 blinks | 0.33 (1.25) | 0.66 (1.82)
  45 deg/ 60 sec | 0.45 (1.45) | 0.63 (1.78)

65. Primary Outcome: Lens Surface Deposits
Description: Assessment of lens front surface deposits. Collected at 2 weeks wear for each lens. (Front surface deposits observed, 0-4, 0=clean, 4=deposits ≥0.5)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
units on a scale | 0.26 (0.31) | 0.41 (0.36)

66. Primary Outcome: Lens Surface Deposits
Description: Assessment of lens front surface deposits. Collected at 4 weeks wear for each lens. (Front surface deposits observed, 0-4, 0=clean, 4=deposits ≥0.5)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Groups:
- Comfilcon A; Lotrafilcon B: Each subject randomized to wear comfilcon A or lotrafilcon B for one month of daily wear before repeating the schedule for the second pair without a washout period. All subjects wore both lenses. (comfilcon A then lotrafilcon B and/or lotrafilcon B then comfilcon A)
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
units on a scale | 0.41 (0.34) | 0.71 (0.41)

67. Primary Outcome: Centration
Description: Assessment of Lens Fit Performance for centration. Collected at 2 weeks for each lens. Proportion of contact lenses fitted where centration was centered or slightly decentered. (Biomicroscopy)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  centered | 94 | 78
  slightly decentered | 6 | 22

68. Primary Outcome: Centration
Description: Assessment of Lens Fit Performance for centration. Collected at 4 weeks for each lens. Proportion of contact lenses fitted where centration was centered or slightly decentered. (Biomicroscopy)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  centered | 93 | 81
  slightly decentered | 7 | 19

69. Primary Outcome: Corneal Coverage
Description: Assessment of Lens Fit Performance for corneal coverage. Collected at 2 weks for each lens. Corneal coverage assessed in primary gaze: (yes=full corneal coverage at all times, no=incomplete corneal coverage)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses | 100 | 100

70. Primary Outcome: Corneal Coverage
Description: Assessment of Lens Fit Performance for corneal coverage. Collected at 4 weeks for each lens. Corneal coverage assessed in primary gaze: (yes=full corneal coverage at all times, no=incomplete corneal coverage)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses | 100 | 100

71. Primary Outcome: Post Blink Movement
Description: Assessment of Lens Fit Performance for post blink movement. Collected at 2 weeks for each lens. (0-4, 0.5 increments; 0=Insufficient, unacceptable movement, 4= Excessive, unacceptable movement)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
units on a scale | 0 (0) | 0.05 (0.22)

72. Primary Outcome: Post Blink Movement
Description: Assessment of Lens Fit Performance for post blink movement. Collected at 4 weeks for each lens. (0-4, 0.5 increments; 0=Insufficient, unacceptable movement, 4= Excessive, unacceptable movement)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
units on a scale | 0.01 (0.09) | 0.05 (0.22)

73. Primary Outcome: Lens Marking Visibility
Description: Assessment of Lens Fit Performance for lens marking visibility. Collected at 2 weeks for each lens. (1-3, 1=excellent, 2=average, 3=poor)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  Excellent | 88 | 27
  Average | 12 | 49
  Poor | 0 | 24

74. Primary Outcome: Lens Marking Visibility
Description: Assessment of Lens Fit Performance for lens marking visibility. Collected at 4 weeks for each lens. (1-3, 1=excellent, 2=average, 3=poor)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  Excellent | 84 | 20
  Average | 16 | 50
  Poor | 0 | 30

75. Primary Outcome: Lens Stability on Blink
Description: Assessment of Lens Fit Performance for lens rotational stability on blink. Collected at 2 weeks for each lens. (No rotation and 5-10 degrees rotation from axis location mark)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  No rotation | 98 | 99
  5-10 degrees | 2 | 1

76. Primary Outcome: Lens Stability on Blink
Description: Assessment of Lens Fit Performance for lens rotational stability on blink. Collected at 4 weeks for each lens. (No rotation and 5-10 degrees rotation from axis location mark)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (lenses) | 120 | 120
percentage of lenses
  No rotation | 100 | 99
  5-10 degrees | 0 | 1

77. Primary Outcome: Lens Stability 5-10 Min
Description: Assessment of Lens Fit Performance for lens to stabilize in 5-10 min. Collected at 2 weeks for each lens. Varied less than 5 degrees from lens marking location between 5-10 min.
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses | 100 | 100

78. Primary Outcome: Lens Stability 5-10 Min
Description: Assessment of Lens Fit Performance for lens to stabilize in 5-10 min. Collected at 4 weeks for each lens. Varied less than 5 degrees from lens marking location between 5-10 min.
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses | 100 | 100

79. Secondary Outcome: Limbal Hyperaemia
Description: Assessment of ocular health. Collected at 2 weeks after removal of lenses. Proportion of eyes with grades 0-1 (No eyes graded >1) (Biomicroscopy, 0-4, ½ grades; 0=none: no injection present, 4=severe)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 99 | 100
  Grade 1/2 | 1 | 0
  Grade 1 | 0 | 0

80. Secondary Outcome: Limbal Hyperaemia
Description: Assessment of ocular health. Collected at 4 weeks after removal of lenses. Proportion of eyes with grades 0-1 (No eyes graded >1) (Biomicroscopy, 0-4, ½ grades; 0=none: no injection present, 4=severe)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 98 | 98
  Grade 1/2 | 2 | 2
  Grade 1 | 0 | 0

81. Secondary Outcome: Bulbar Hyperaemia
Description: as for outcome 2
Time Frame: Baseline
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Overall Study Group: All 60 subjects with habitual lens prior to dispense of study lens.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 98.4
  Grade 1/2 | 1.6
  Grade 1 | 0.0

82. Secondary Outcome: Bulbar Hyperaemia
Description: as for outcome 79
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 95
  Grade 1/2 | 0 | 5
  Grade 1 | 0 | 0

83. Secondary Outcome: Bulbar Hyperaemia
Description: as for outcome 80
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 94
  Grade 1/2 | 0 | 6
  Grade 1 | 0 | 0

84. Secondary Outcome: Lower Palpebral Hyperaemia
Description: as for outcome 2
Time Frame: Baseline
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 92.5
  Grade 1/2 | 7.5
  Grade 1 | 0.0

85. Secondary Outcome: Lower Palpebral Hyperaemia
Description: as for outcome 79
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 96 | 82
  Grade 1/2 | 4 | 18
  Grade 1 | 0 | 0

86. Secondary Outcome: Lower Palpebral Hyperaemia
Description: as for outcome 80
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 93 | 78
  Grade 1/2 | 7 | 20
  Grade 1 | 0 | 2

87. Secondary Outcome: Corneal Stromal Haze
Description: as for outcome 2
Time Frame: Baseline
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 100
  Grade 1/2 | 0.0
  Grade 1 | 0.0

88. Secondary Outcome: Corneal Stromal Haze
Description: as for outcome 79
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 100
  Grade 1/2 | 0 | 0
  Grade 1 | 0 | 0

89. Secondary Outcome: Corneal Stromal Haze
Description: as for outcome 80
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 100
  Grade 1/2 | 0 | 0
  Grade 1 | 0 | 0

90. Secondary Outcome: Corneal Neovascularization
Description: Investigators' objective assessment of ocular health. Collected at baseline after removal of habitual lenses. Proportion of eyes with grades 0-1 (No eyes graded >1) (Biomicroscopy, 0-4, ½ grades; 0=none: no injection present, 4=severe)
Time Frame: Baseline
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 96.7
  Grade 1/2 | 3.3
  Grade 1 | 0.0

91. Secondary Outcome: Corneal Neovascularization
Description: as for outcome 79
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 96
  Grade 1/2 | 0 | 4
  Grade 1 | 0 | 0

92. Secondary Outcome: Corneal Neovascularization
Description: as for outcome 80
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 97
  Grade 1/2 | 0 | 3
  Grade 1 | 0 | 0

93. Primary Outcome: Overall Stability
Description: Assessment of Lens Fit Performance for overall lens stability. Collected at 2 weeks for each lens. (Excellent or Good.
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Excellent | 74 | 38
  Good | 26 | 62

94. Primary Outcome: Overall Stability
Description: Assessment of Lens Fit Performance for overall lens stability. Collected at 4 weeks for each lens. (Excellent or Good.
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Excellent | 72 | 36
  Good | 28 | 64

95. Primary Outcome: Overall Fit Acceptance
Description: Assessment of Lens Fit Performance for overall lens fit acceptance. Collected at 2 weeks for each lens. Rated perfect or not perfect based on lens fit alone. (0-4; 0=should not be worn, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Perfect | 76 | 49
  Not Perfect | 24 | 51

96. Primary Outcome: Overall Fit Acceptance
Description: Assessment of Lens Fit Performance for overall lens fit acceptance. Collected at 4 weeks for each lens. Rated perfect or not perfect based on lens fit alone. (0-4; 0=should not be worn, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Lenses) | 120 | 120
percentage of lenses
  Perfect | 73 | 44
  Not Perfect | 27 | 56

97. Secondary Outcome: Corneal Infiltrates
Description: as for outcome 2
Time Frame: Baseline
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
percentage of eyes
  Grade 0 | 100
  Grade 1/2 | 0.0
  Grade 1 | 0.0

98. Secondary Outcome: Corneal Infiltrates
Description: as for outcome 79
Time Frame: 2 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 100
  Grade 1/2 | 0 | 0
  Grade 1 | 0 | 0

99. Secondary Outcome: Corneal Infiltrates
Description: as for outcome 80
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Grade 0 | 100 | 100
  Grade 1/2 | 0 | 0
  Grade 1 | 0 | 0

100. Secondary Outcome: Participant Preference for Their Habitual Lenses or the First Study Lenses (Lotrafilcon B)
Description: Participant preference for their habitual lenses or the first study lenses during the last two weeks with regard to comfort, dryness, handling, vision, lens fit and overall. (Forced choice; habitual, study lenses)
Time Frame: 2 weeks
Population: All 60 subjects were habitual lense wearers and randomized to both sets of study lenses.
Measure: Number; unit: percentage of patients
Groups:
- Habitual Lenses; Lotrafilcon B: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
Arm/Group | Habitual Lenses | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of patients
  Comfort | 55 | 45
  Dryness | 57 | 43
  Handling | 55 | 45
  Vision | 47 | 53
  Lens Fit | 43 | 57
  Overall | 53 | 47

101. Secondary Outcome: Participant Preference for Their Habitual Lenses or the First Study Lenses (Comfilcon A)
Description: as for outcome 100
Time Frame: 2 weeks
Population: All 60 subjects were habitual lense wearers and randomized to both sets of study lenses.
Measure: Number; unit: percentage of patients
Arm/Group | Habitual Lenses | Comfilcon A
Number analyzed (Participants) | 60 | 60
percentage of patients
  Comfort | 20 | 80
  Dryness | 18 | 82
  Handling | 55 | 45
  Vision | 25 | 75
  Lens Fit | 30 | 70
  Overall | 25 | 75

102. Secondary Outcome: Participant Preference for Their Habitual Lenses or the First Study Lenses (Lotrafilcon B)
Description: Participant preference for their habitual lenses or the first study lenses during the last four weeks with regard to comfort, dryness, handling, vision, lens fit and overall. (Forced choice; habitual, study lenses)
Time Frame: 4 weeks
Population: All 60 subjects were habitual lense wearers and randomized to both sets of study lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lenses | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Comfort | 62 | 38
  Dryness | 58 | 42
  Handling | 57 | 43
  Vision | 45 | 55
  Lens Fit | 52 | 48
  Overall | 55 | 45

103. Secondary Outcome: Participant Preference for Their Habitual Lenses or the First Study Lenses (Comfilcon A)
Description: as for outcome 102
Time Frame: 4 weeks
Population: All 60 subjects were habitual lense wearers and randomized to both sets of study lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Habitual Lenses | Comfilcon A
Number analyzed (Participants) | 60 | 60
percentage of participants
  Comfort | 20 | 80
  Dryness | 22 | 78
  Handling | 52 | 48
  Vision | 27 | 73
  Lens Fit | 27 | 73
  Overall | 23 | 77

104. Secondary Outcome: Participants Likelihood of Switching From Habitual Lenses to the Study Lenses
Description: Participants likelihood of switching from habitual lenses to either pair of the study lenses when asked; How likely are they to switch from their habitual lenses to either the first study lenses or the second study lenses?" Collected at 4 weeks for each study pair. (4 point Likert scale; very likely, likely, unlikely, very unlikely)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of particpants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of particpants
  Very Likely | 45 | 10
  Likely | 32 | 32
  Unlikely | 22 | 42
  Very Unlikely | 2 | 17

105. Secondary Outcome: Participants Likelihood of Continuing to Wear the Study Lenses.
Description: Participants likelihood of continuing to wear either of the pairs of study lenses when asked; "How likely are they to continue to wearing either the first study lenses or the second study lenses?" Collected at 4 weeks fore each study pair. (4 point Likert scale; very likely, likely, unlikely, very unlikely)
Time Frame: 4 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Very Likely | 45 | 12
  Likely | 32 | 30
  Unlikely | 22 | 42
  Very Unlikely | 2 | 17

106. Secondary Outcome: Participant Recommendation of a Study Lens to Friends, Family or Colleagues
Description: Percentage of participants that answer the question, "What study lens they will most likely recommend to friends, family or colleagues?" Collected at end of study. (Forced choice; First Study Lenses, Second Study Lenses)
Time Frame: 8 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants | 77 | 23

107. Secondary Outcome: Participant Likelihood of Recommending a Study Lens to Friends, Family or Colleagues.
Description: Percentage of participants that answer the question, "How likely are they to recommend either the first pair of study lenses or the second pair of study lenses to friends, family or colleagues?" Collected at study end. (4 point Likert scale; very likely, likely, unlikely, very unlikely)
Time Frame: 8 weeks
Population: All 60 subjects randomized to both sets of lenses.
Measure: Number; unit: percentage of participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 60
percentage of participants
  Very Likely | 52 | 15
  Likely | 35 | 40
  Unlikely | 11 | 35
  Very Unlikely | 2 | 10

108. Secondary Outcome: Participant Preference for Their Habitual Lenses or Either of the Study Lenses
Description: Percentage of participants that answer the question, "Which type of study lens they prefer with regard to comfort, dryness, handling, vision, lens fit and overall performance?" Collected at study end. (Forced choice; habitual lenses, first study lenses, second study lenses)
Time Frame: 8 weeks
Population: All 60 subjects wore habitual lenses prior to randomization of study lenses.
Measure: Number; unit: percentage of participants
Groups:
- Habitual: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
Arm/Group | Comfilcon A | Lotrafilcon B | Habitual
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants
  Comfort | 72 | 15 | 13
  Dryness | 68 | 17 | 15
  Handling | 27 | 42 | 31
  Lens Fit | 47 | 42 | 11
  Vision | 60 | 30 | 10
  Overall | 65 | 23 | 12

109. Secondary Outcome: Participant Preference for Either of the Study Lenses
Description: Percentage of participants that answer the question, "Which type of study lens they prefer with regard to comfort, dryness, handling, vision, lens fit and overall performance?" Collected at study end. (Forced choice; first study lenses, second study lenses, neither)
Time Frame: 8 weeks
Population: All 60 subjects wore habitual lenses prior to randomization of study lenses.
Measure: Number; unit: percentage of participants
Groups:
- Neither: All subjects were habitual lens wearers and were randomized to a pair of study lenses. All wore the study lenses for a minimum of 8 hours a day, 7 days a week and one month of daily wear before repeating the schedule for the second pair without a washout period.
Arm/Group | Comfilcon A | Lotrafilcon B | Neither
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants
  Comfort | 80 | 20 | 0
  Dryness | 80 | 20 | 0
  Handling | 40 | 55 | 5
  Lens Fit | 58 | 38 | 4
  Vision | 70 | 28 | 2
  Overall | 78 | 22 | 0

ADVERSE EVENTS:
Time Frame: From dispense up to one month for each pair of lenses.
Arm/Group | Comfilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.